CLINICAL TRIAL: NCT05525624
Title: Evaluation of the Effectiveness of Transition Model-Based Discharge Training in Parents of Preterm Infants:Double Blinded A Randomized Controlled Study
Brief Title: Transition Model-Based Discharge Training in Parents of Preterm Infants
Acronym: TRAMPRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Serife Tutar, Dr.Şerife Tutar, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0732
Record Dates: First submitted 2022-02-27; First posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-04

CONDITIONS: Preterm Infant; Parents; Premature Birth; Randomized Controlled Trial; Transitional Care
MeSH Terms: conditions — Premature Birth | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Transition Model is discharge model in preterm infants.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The research will be conducted in a double-blind design and the data of the research will be collected by the clinical nurse. Parents participating in the research will not know that they are in the intervention or control group. Telephone support during the research process will be provided by an independent interviewer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): TRAMPRE is an acronym that defines multimodal interventions discharge training. TRAMPRE will be applied to the participants in line with the "Preterm Baby Care Guide" at the discharge stage. Weekly telephone follow-up will be carried out for 12 weeks after discharge. Applications to be made to the initiative group are given below. Phone Follow-up/Interview: During the first 12 weeks following the discharge of the preterm baby, parents will be interviewed by phone at least once a week.
  Interventions: Device: TRAMPRE
- Control Group (Active Comparator): Participants in this group will be included in the routine neonatal clinic discharge training of the hospital where the research was conducted and no intervention will be applied.
  Interventions: Other: Control Group

INTERVENTIONS:
Device: TRAMPRE — discharge interventions Transition Model is discharge interventions in parents of preterm infants.
  Other Names: discharge interventions
  Arms: Experimental
Other: Control Group — routine neonatal clinic discharge training of the hospital
  Other Names: routine neonatal clinic discharge training
  Arms: Control Group

SUMMARY:
Infant and Child Monitoring Protocol prepared by the General Directorate of Mother and Child Health and Family Planning of the Ministry of Health regarding the monitoring of postpartum processes in our country. However, there is no separate recommendation for home follow-up and care of mothers and babies who gave birth preterm. In addition, there are deficiencies in the effective conduct of home visits specified in these guides. In addition to the parents' lack of knowledge about the long-term follow-up and care of these babies, the coordination between primary and secondary health care providers and senior health care providers is not at the desired level. In addition to all these, services such as training and consultancy cannot be carried out due to disruptions in many polyclinic services due to the COVID-19 pandemic worldwide. For this reason, there is a need to develop programs for home care and follow-up of preterm infants, who are a sensitive population, in terms of both reducing the patient density in hospitals and reducing the hospital return rates of preterm infants. In this context, the aim of our research is; The aim of this study is to evaluate the effectiveness of discharge training based on the Transition Model in parents with preterm infants.H1: In the group in which the interventions based on the Transition Model are applied, the information needs of the parents will be met more compared to the control group. H1: Parent-infant role development will be higher in the group in which interventions based on the Transition Model are applied. H1: The level of coping with stress will be better in the group in which interventions based on the Transition Model are applied. H1: The level of grief will be lower in the group in which interventions based on the Transition Model are applied. H1: The level of postpartum depression will be lower in the group in which interventions based on the Transition Model are applied. H1: Babies in the group in which interventions based on the Transition Model are applied will have fewer hospital admissions, except for the planned outpatient visit

DETAILED DESCRIPTION:
Intervention Group: The intervention protocol of the research will be based on the Transition Model. Discharge training will be applied to the participants in line with the "Preterm Baby Care Guide" at the discharge stage. Weekly telephone follow-up will be carried out for 12 weeks after discharge. Applications to be made to the initiative group are given below. Phone Follow-up/Interview: During the first 12 weeks following the discharge of the preterm baby, parents will be interviewed by phone at least once a week. During the interview, issues concerning the baby's health status (baby bed, physical conditions of the house, newborn jaundice, nutrition, etc.) will be included in the scope of the interview and suggestions will be made for the baby's growth and development in healthy conditions (safe sleep, clothing selection, etc.). Interviews will be held in line with the "Baby Care Skill Form" and each interview will be recorded in the form. The duration and number of interviews will be determined according to the needs of the parent. In addition, in this process, information such as which health institution application has been made, the degree of the institution applied (primary / secondary / tertiary health institution) will be recorded. Control Group: Participants in this group will be included in the routine neonatal clinic discharge training of the hospital where the research was conducted and no intervention will be applied. The Parents and Preterm Baby General Information Form will be applied to the parents who agreed to participate in the study at the first interview, and when the data collection process of the research is completed, these parents will be contacted by phone and the Transition Scale and Edinburgh Postnatal Depression Scale will be applied. As in the intervention group, information such as the status of application to the health institution, the reason for the application and the degree of the institution applied to (primary / secondary / tertiary health institution) will be recorded in this group. Statistical Package of Social Science (SPSS 23) package program will be used in the evaluation of the data obtained from the research. For the intervention and control groups, the Cronbach Alpha coefficient, scale score average and minimum-maximum values will be calculated for the pre-test and post-test. In order to compare the pre-test and post-test data of the intervention and control groups, the t-test for the difference of the mean of the two peer groups (t-test of two paired groups), the Wilcoxon Signed Ranks Test, and the Wilcoxon Signed Ranks Test, and the Mann Whitney-U Test for the data without normal distribution will be performed.

ELIGIBILITY:
Inclusion Criteria:

* For mothers;

  * Having given birth between 340/7-366/7 weeks
  * Absence of a chronic disease that may affect physical and mental care
  * Residing within the provincial borders of Antalya
* For babies;

  * No congenital anomalies
  * Postpartum neonatal asphyxia, respiratory distress syndrome, intraventricular hemorrhage and necrotizing enterocolitis etc. no problem
  * Postpartum Apgar score >7 Babies discharged after being followed up in
  * The neonatal clinic will be included in the study

Exclusion Criteria:

* For mothers;

  *Having a physical or mental chronic illness that may affect the baby's care process
* For babies;

  * Neonatal asphyxia, respiratory distress syndrome, intraventricular hemorrhage and necrotizing enterocolitis etc. receiving ventilator support after delivery.
  * Babies with a problem will not be included in the study.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Mothers of preterm infants were included in the study because mothers are involved in primary infant care
Enrollment: 200 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Effect of TRAMPRE | Change from baseline effect of TRAMPRE at 3 months
  TRAMPRE will be applied to the participants in line with the "Preterm Baby Care Guide" at the discharge stage. Weekly telephone follow-up will be carried out for 12 weeks after discharge. Applications to be made to the initiative group are given below. Phone Follow-up/Interview: During the first 12 weeks following the discharge of the preterm baby, parents will be interviewed by phone at least once a week.

SECONDARY OUTCOMES:
Level of postpartum depression | Change from baseline level of postpartum depression at 3 months
  The Edinburgh Postpartum Depression Scale will be administered three months after discharge.
Frequency of readmission | Change from baseline Frequency of readmission at 3 months
  Planned/unplanned admission to hospital after discharge:It is planned to be used in weekly planned parent interviews after discharge. The content of the form includes questions about hospital applications after discharge and the reasons for application.

CONTACTS AND LOCATIONS:
Overall Officials: Şerife Tutar, Principal Investigator — Suleyman Demirel University
Locations (2):
- Turkey (Türkiye) (2):
  - Suleyman Demirel University, Isparta
  - Şerife Tutar, Isparta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tutar S, Demir Avci Y, Gozum S. The Effect of Transition Model-Based Discharge Training for Mothers of Late Preterm Infants (TRAMPRE): A Randomized Controlled Study. Res Nurs Health. 2025 Dec;48(6):692-705. doi: 10.1002/nur.70017. Epub 2025 Aug 23. PMID 40847827